CLINICAL TRIAL: NCT03866083
Title: Safety and Efficacy of Extracorporeal Cytokine Hemoadsorption in Septic Shock in Critically Ill Cirrhotics -A Prospective Randomized Controlled Trial
Brief Title: Safety and Efficacy of Extracorporeal Cytokine Hemoadsorption in Septic Shock in Critically Ill Cirrhotics
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-Sepsis-20
Record Dates: First submitted 2019-03-04; First posted 2019-03-07 (Actual); Last update posted 2019-05-01 (Actual); Status verified 2019-03

CONDITIONS: Septic Shock
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Extracorporeal Cytokine hemadsorption therapy (Experimental): Hemoperfusion will be carried out for one session within 12 hours for all randomized patient using the adsorption columns for Jianfan Biotechnology Co., Zhuhai, China). The hemoperfusion apparatus will be connected in front of the hemodialyzer in series.
  Interventions: Drug: Extracorporeal Cytokine hemadsorption therapy; Drug: Standard Medical Treatment
- Stadard Medical treatment (Active Comparator): Stadard Medical treatment
  Interventions: Drug: Standard Medical Treatment

INTERVENTIONS:
Drug: Extracorporeal Cytokine hemadsorption therapy — Hemoperfusion will be carried out for one session within 12 hours for all randomized patient using the adsorption columns for Jianfan Biotechnology Co., Zhuhai, China). The hemoperfusion apparatus will be connected in front of the hemodialyzer in series.
  Arms: Extracorporeal Cytokine hemadsorption therapy
Drug: Standard Medical Treatment — Standard Medical Treatment

SUMMARY:
Patients with septic shock would be screened. Following this, patients meeting the inclusion and exclusion criteria will be screened and randomized to the two treatment groups. Standard criteria will be considered to define refractoriness to fluids. In all patients, baseline endotoxin activity assay and blood and urine sample will be stored for looking at the effect of therapy on these factors. Septic shock would be defined as clinical construct of sepsis with persisting hypotension requiring vasopressors to maintain MAP>=65 mm of Hg and having a serum lactate >2 mmol/L despite adequate volume resuscitation. Patients assigned to the treatment arm and who do not already have access for dialysis will have a standard hemodialysis catheter inserted in one of the femoral veins by the physician. Hemoperfusion will be carried out for one session within 12 hours for all randomized patient using the adsorption columns for Jianfan Biotechnology Co., Zhuhai, China). The hemoperfusion apparatus will be connected in front of the hemodialyzer in series. The procedure would be done for 2 hours without use of heparin with use of normal saline for pipeline flushing. In patients who also require hemodialysis the dialysis would subsequently be continued. Subsequent sessions of therapy would be done for patients (if required).

ELIGIBILITY:
Inclusion Criteria:

- Critically ill cirrhotics with early onset septic shock (<24 hours) with norepinephrine of more than 10 ug/min and lactate >4 mmol/L.

Exclusion Criteria:

* Patients with age less than 18 years
* Severe known cardiopulmonary disease (structural or valvular heart disease, coronary artery disease, COPD)
* Severe coagulopathy platelets <20,000 and INR >5
* Active Bleed (Mucosal or variceal)
* Pregnancy
* Chronic kidney disease
* Extremely moribund patients with an expected life expectancy of less than 24 hours
* Failure to give informed consent from family members.
* Hemodynamic instability requiring very high dose of vasopressors, late presentation or spontaneous reversal of shock
* Patient enrolled in other clinical trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-06-30 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
Reversal of shock in both groups | 72 hours

SECONDARY OUTCOMES:
Mortality in both groups | 28 days
Duration of mechanical ventilation in both groups | 3 months
Number of days in Intensive Care Unit stay in both groups | 3 months
Reversal of Acute Kidney Injury | 5 days
Lactate clearance in both groups | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver & Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided